CLINICAL TRIAL: NCT00242879
Title: Phase IIB, Randomized, Multicenter, Parallel Group, Study to Evaluate the Safety, Pharmacokinetics and Antiviral Effect of Four Blinded Dosing Regimens of GW640385X/Ritonavir Compared to Open-label Current PI Therapy in HIV-1 Infected, Protease Inhibitor Experienced Adults for 2 Weeks With Long-term Assessment (>48 Weeks) of Safety, Pharmacokinetic and Antiviral Activity of Selected 385/RTV Dosing Regimen(s) vs. a Ritonavir-boosted, Protease Inhibitor Containing Regimen
Brief Title: A Dose Ranging Study Of GW640385 Boosted With Ritonavir (Rtv) In Comparison To A RTV-Boosted Protease Inhibitor (PI) In HIV-1 Infected PI-Experienced Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPR20001
Record Dates: First submitted 2005-10-19; First posted 2005-10-21 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Infection, Human Immunodeficiency Virus I; HIV-1 Infection
Keywords: treatment-experienced; RTV; protease inhibitor; ritonavir; GW640385; HIV-1
MeSH Terms: conditions — Infections | interventions — Ritonavir

INTERVENTIONS:
Drug: Physician determined comparator PI + ritonavir
Drug: GW640385 + ritonavir
  Other Names: Physician determined comparator PI + ritonavir

SUMMARY:
This is a two phase study (randomised and non-randomised phase). The randomised phase will initially examine 4 blinded doses of GW640385 boosted with rtv (with continuation of current background therapy) in comparison to an ongoing, open-labeled rtv-boosted protease inhibitor (PI) regimen for 15 days. At the Day 15 visit, all subjects will optimize background therapy. Additionally, subjects receiving the lowest dose of GW640385 will be re-randomised to one of the higher doses and subjects in the control arm will receive a new rtv-boosted PI based on resistance testing at screening. Subjects will remain in the randomized phase on one of these 4 continuing treatment arms for at least 48 weeks. An interim analysis will occur during the randomised phase to select for a dose of GW640385 to evaluate further in Phase III studies. After dose selection subjects will move to the non-randomised phase of the study. In the non-randomised phase subjects who are receiving GW640385 will be assigned to final selected dose for assessment of long term safety, tolerability, pharmacokinetics, and antiviral activity.

DETAILED DESCRIPTION:
A Phase IIB, Randomized, Multicenter, Parallel Group Study to Evaluate the Short-Term Safety, PK and Antiviral Activity of Four Dosing Regimens of GW640385/rtv Therapy Compared to Open-label Current Protease Inhibitor (PI) Therapy in HIV-1, PI-Experienced Adults for 2 wks with Long-Term Evaluation (>48 wks) of Safety, PK and Antiviral Activity of Selected GW640385/rtv Dosing Regimen(s) vs. a RTV-boosted, PI Containing Regimen

ELIGIBILITY:
Inclusion criteria:

* 18+ years of age (or =16 years of age for non-EU countries, according to local requirements).
* HIV-1 infected subjects.
* Females must be of either non-childbearing potential or have a negative pregnancy test at Screening and agree to use a protocol approved method of contraception.
* Plasma HIV-1 RNA (viral load) =1,000 copies/mL at Screening.
* Evidence of at least 2 multi-PI resistant mutations at Screening or within 3 months of Screening.
* Subjects must have been receiving the same anti-HIV medicines that they are on currently for at least 8 weeks prior to Screening; these anti-HIV medicines will include a single protease inhibitor (PI) in combination with a low dose of ritonavir (i.e., a ritonavir-boosted PI). However, the current PI cannot be tipranavir.
* Able to understand and follow protocol requirements, instructions and protocol-stated restrictions.
* Be willing and able to provide signed and dated written informed consent prior to study entry.

Exclusion criteria:

* Subjects cannot change their anti-HIV medicines between Screening and Day 1 Visit.
* Subjects can not be receiving dual ritonavir-boosted PIs, non-nucleoside reverse transcriptase inhibitors (NNRTIs) or Tipranavir at Screening.
* Active CDC Class C disease at screening.
* Pregnant or breastfeeding women.
* Protocol-specified laboratory abnormalities at Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2005-08; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Time averaged change in plasma HIV-1 RNA over 16 wks
Proportion of subjects achieving the target pharmacokinetic (PK) GW640385 drug levels
Change in laboratory parameters

SECONDARY OUTCOMES:
Assessments of HIV viral load changes
GW640385 and RTV pharmacokinetic measurements
The incidence of adverse events
Changes in laboratory measurements
ECG measurements
HIV viral resistance assessment
Immunologic measures

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (57):
- United States (23):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Norwalk, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Bradenton, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Miami Beach, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Hampton, Virginia
- Australia (3):
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Liverpool, New South Wales
  - GSK Investigational Site, South Yarra, Victoria
- GSK Investigational Site, Brussels, Belgium
- Canada (4):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
- France (5):
  - GSK Investigational Site, Caen
  - GSK Investigational Site, La Roche-sur-Yon
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
- Germany (6):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Italy (7):
  - GSK Investigational Site, Bari, Apulia
  - GSK Investigational Site, Ferrara, Emilia-Romagna
  - GSK Investigational Site, Rimini, Emilia-Romagna
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Bagno A Ripoli (FI), Tuscany
- Portugal (2):
  - GSK Investigational Site, Cascais
  - GSK Investigational Site, Lisbon
- Puerto Rico (2):
  - GSK Investigational Site, Ponce
  - GSK Investigational Site, San Juan
- Romania (3):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Constanța
  - GSK Investigational Site, Iași
- GSK Investigational Site, London, United Kingdom